CLINICAL TRIAL: NCT06264115
Title: Outcomes of Three Ports Versus Four Ports Laparoscopic Cholecystectomy, Sohag General Surgery Department Experience
Status: Enrolling by invitation | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mikel Mokhtar Shafik, Resident of general surgery of sohag university hospital, Sohag University
Other Study IDs: Soh-Med-24-01-05MS
Record Dates: First submitted 2024-02-01; First posted 2024-02-16 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Cholecystitis, Chronic
MeSH Terms: conditions — Cholecystitis; Bronchiolitis Obliterans Syndrome | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Three ports Laparoscopic Cholecystectomy group
  Interventions: Procedure: Laparoscopic Cholecystectomy
- Four ports Laparoscopic Cholecystectomy group
  Interventions: Procedure: Laparoscopic Cholecystectomy

INTERVENTIONS:
Procedure: Laparoscopic Cholecystectomy — Using Three Ports or Four Ports for Laparoscopic Cholecystectomy

SUMMARY:
To compare the outcomes of three ports and four ports Laparoscopic Cholecystectomy

DETAILED DESCRIPTION:
To compare the outcomes of three ports and four ports Laparoscopic Cholecystectomy Randomized clinical trial comparative study will be carried out on 50 patients underwent laparoscopic cholecystectomy in general surgical department, Sohag University. An informed written consent will be obtained from the patients. Every patient will receive an explanation of the purpose of the study and will have a secret code number. Research results will be only used for scientific purposes. Any unexpected risks appearing during the course of research will be clarified to the participants and to the ethical committee on time.

Patients will be randomly classified into two equal groups; 25 patients will be enrolled in each group using computer generated random number in closed sealed envelope.

Group I (3-ports): 25 patients undergo a three-port LC. Group II (4-ports): 25 patients undergo a four-port LC. All patients will be subjected to thorough history taking (age, sex, symptoms, and duration of symptoms) and full clinical evaluation.

Abdominal ultrasound will be done in all patients. Baseline laboratory (complete blood count and coagulation profile) will be ordered in all patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years.
* Both sexes.
* Patient with clinical, laboratory and/or radiological evidence that is a candidate for cholecystectomy operation.

Exclusion Criteria:

* Patient's refusal.
* Bile duct stones.
* History of obstructive jaundice.
* Severe acute calculus pancreatitis.
* Severe co-morbid diseases (uncontrolled diabetes, hypertension, and severe direct hyperbilirubinemia).
* Prior surgery or adhesion.
* Radical cholecystectomy.
* Pregnancy.
* Malignancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients undergoing laparoscopic cholecystectomy
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain score | One year
  Measurement of postoperative pain in both groups according to visual analogue scale The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').
  Ask the patient to rate their current level of pain by placing a mark on the line. Use a ruler to measure the distance in centimetres from the 'no pain marker' (or zero) to the current pain mark. This provides a pain intensity score out of 10; for example, 6 out of 10 (or 6/10).

SECONDARY OUTCOMES:
Operative time | One year
length of hospital stay | one year

OTHER OUTCOMES:
Total postoperative morphine consumption | one year
Time of first analgesic | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university, Sohag, Egypt